CLINICAL TRIAL: NCT05238038
Title: Electrical Impedance Tomography for the Assessment of Neurological Disease
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Seward Rutkove, Chairman, Department of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2019P000431
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Neuromuscular Disease Patients; Central Neurological Disease Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: EIT measurements will be performed on appendicular muscles (in the upper and lower extremities) depending on the condition, both at rest and with contraction. EIT measurements will be repeated on an intermittent basis to assess repeatability as well disease progression or improvement over time
- Neuromuscular disease patients and Central neurological disease patients: EIT measurements will be performed on appendicular muscles (in the upper and lower extremities) depending on the condition, both at rest and with contraction. EIT measurements will be repeated on an intermittent basis to assess repeatability as well disease progression or improvement over time

SUMMARY:
Overview of study. This is an observational study that is intended to provide the first in-human data using EIT as a biomarker of muscle health in neuromuscular conditions. We will seek patients with neurological disorders (both neuromuscular and other neurological conditions) as well as healthy subjects for study. EIT measurements will be performed on appendicular muscles (in the upper and lower extremities) depending on the condition, both at rest and with contraction. EIT measurements will be repeated on an intermittent basis to assess repeatability as well disease progression or improvement over time.

DETAILED DESCRIPTION:
1. Overview of study. This is an observational study that is intended to provide the first in-human data using EIT as a biomarker of muscle health in neuromuscular conditions. We will seek patients with neurological disorders (both neuromuscular and other neurological conditions) as well as healthy subjects for study. EIT measurements will be performed on appendicular muscles (in the upper and lower extremities) depending on the condition, both at rest and with contraction. EIT measurements will be repeated on an intermittent basis to assess repeatability as well disease progression or improvement over time.
2. History and examination (All participants). After reviewing the purpose and procedures of the study, the subject, or a legally authorized representative (LAR), will be asked to sign the internal review board-approved informed consent form.

   Basic medical, social, and family histories will then be obtained and recorded. Previous medical records will be reviewed and the neurological diagnosis confirmed when possible. Information including Body Mass Index (BMI), presence of a gastrostomy, imaging findings, and blood tests will be noted when available. Medications, including drug doses, history of recent medication changes, and duration of treatment) will be reviewed.

   Brief general neurological examinations will then be completed.
3. EIT measurements (All participants).We will be using a SwissTom Pioneer EIT data acquisition system. SwissTom has developed a clinical EIT system which is not FDA-approved, although approved in Europe for lung imaging. It comprises an elastic belt that is connected to a computer via a universal serial bus (USB) or an Ethernet cable. Via multiple surface electrodes on the belt, EIT data is captured and transmitted via the USB or Ethernet cable to the computer. Low resolution, tomography-like impedance images of the muscle are computed and displayed on the computer. The impedance images will be used to evaluate muscle recruitment and other muscle function parameters.

   The data acquisition system includes a unit that transmits a small imperceptible electrical current into the chest, via a pair of operator-selected electrodes, while voltage is sensed on all remaining electrodes. The frequency of the transmitted current ranges from 100 Hz to 1 MHz. For frequencies from 100 Hz to 1 kHz, the current amplitude is limited to a maximum of 0.1 mA. From 1 kHz to 100 kHz, the current amplitude is limited to a maximum of 0.1*f mA, where f is the frequency of the current. For frequencies higher than 100 kHz, the current amplitude is limited to a maximum of 10 mA. This meets the safety requirements for applied current as specified in the International Electrotechnical Commission (IEC) 60601-1 safety standard for medical devices.

   During data acquisition, the patient may be asked to contract the muscles against resistance of the examiner or against a standard force transducer. The patient may also be asked to contract the muscle while holding a weight in the hand or with a weighted band around the ankle.

   EIT measurements may be repeated to assess repeatability within the session.
4. Ultrasound measurements. An FDA-approved Terason t3000 system may be performed on the muscle or muscle region being assessed in order to better assess the internal anatomy of the region being imaged. These measurements may be done with muscle in a relaxed or a contracted state depending on the specific situation.
5. Handheld dynamometry. In patients who have weakness on standard neurological examination, further quantification of weakness may be obtained by performing handheld dynamometry using a MicroFet2 handheld dynamometry (Hoggan Health Industries, Provo, UT) on relevant muscles. A trained examiner may perform all measurements and the best of 3 trials utilized.
6. Relevant validated questionnaires. Depending on the disease, appropriate validated scales may be incorporated including the amyotrophic lateral sclerosis functional rating scale-revised (ALSFRS-R, ALS patients only) or the Unified Parkinson's Disease Rating Scale (UPDRS, Parkinson's Disease patients only).
7. Follow-up visits. Depending on the diagnosis, the participant will be asked if they are willing to return for follow-up at some later point (likely 3-months to 1-year later, depending the specific diagnosis and subject convenience).

ELIGIBILITY:
Healthy volunteers

Inclusion Criteria:

* Age 21 to 80 years

Exclusion Criteria:

* Generalized neuromuscular disease or debilitated state due to underlying medical disease such as heart failure or malignancy

Neuromuscular disease patients:

Inclusion criteria:

1. Age 21 to 80 years;
2. History of awell-defined, localized or generalized neuromuscular condition producing weakness or muscle atrophy, including disuse atrophy.

Exclusion criteria:

1. Multiple generalized neuromuscular conditions.

Central neurological disease patients:

Inclusion criteria:

1. Age 21 to 80 years;
2. History of a well-defined disorder affecting the central nervous system that impacts motor function, including stroke, Parkinson's disease, dystonia, and multiple sclerosis

Exclusion criteria:

1. Multiple generalized neuromuscular conditions.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neuromuscular disease patients (well-defined, localized or generalized neuromuscular condition producing weakness or muscle atrophy, including disuse atrophy) and Central neurological disease patients (well-defined disorder affecting the central nervous system that impacts motor function, including stroke, Parkinson's disease, dystonia, and multiple sclerosis)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
To establish normative values for EIT data and reproducibility in adult healthy subjects. | 1 year
  First, we will assess simple percent variability by comparing test-retest measurements and calculating absolute value differences. Secondly, we will perform intraclass correlation analysis of test-retest data. Third, we will perform Bland-Altman analyses with calculation of precision. By performing all three approaches, we will obtain the most complete assessment of the technique's reliability.

SECONDARY OUTCOMES:
To identify EIT signal data to assist in characterizing muscle as impacted by neuromuscular diseases versus healthy controls versus central neurological conditions. | 1 year
  We will test for over-fitting the data and ensure that the outcomes used are generally applicable. Initial analysis will consist of one-way ANOVA with post-hoc t-tests to confirm basic discrimination followed by ROC analyses. The goal will be to identify the best set of metrics for disease discrimination.

CONTACTS AND LOCATIONS:
Overall Officials: Seward Rutkove, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States